CLINICAL TRIAL: NCT01346774
Title: Phase II Efficacy of Cranberry Powder in Preventing Catheter-associated Urinary Tract Infection Post Elective Gynecological Surgery
Brief Title: Preventing Urinary Tract Infection Post-Surgery
Acronym: PUPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Betsy Foxman (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Michigan (Other)
Responsible Party: Sponsor-Investigator, Betsy Foxman, Hunein F & Hilda Maassab Professor of Epidemiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R21DK085290 (NIH); HUM00041108 (Other: University of Michigan IRBMED); R21DK085290 (NIH)
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Urinary Tract Infection
Keywords: cystitis; pyelonephritis; bladder infection; kidney infection
MeSH Terms: conditions — Urinary Tract Infections; Cystitis; Pyelonephritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cranberry powder capsules (Experimental): TheraCran® cranberry: based upon proanthocyanidin content, the four cranberry capsules are equivalent to two 8-ounce servings of cranberry juice.
  Participants were directed to take two capsules by mouth twice each day (once in the morning and once in the evening) starting at time of discharge for 4-6 weeks, or until their return for their post-operative doctor's visit. Participants were instructed to drink an 8 oz glass of water while taking the capsule with or without food.
  Interventions: Drug: Cranberry powder capsules
- Placebo capsules (Placebo Comparator): Placebo: participants were directed to take two capsules by mouth twice each day (once in the morning and once in the evening) starting at time of discharge for 4-6 weeks, or until their return for their post-operative doctor's visit. Participants were instructed to drink an 8 oz glass of water while taking the capsule with or without food.
  Interventions: Drug: Placebo powder capsules

INTERVENTIONS:
Drug: Cranberry powder capsules — 2 cranberry powder capsules twice a day
  Other Names: TheraCran
  Arms: Cranberry powder capsules
Drug: Placebo powder capsules — 2 placebo capsules twice a day
  Arms: Placebo capsules

SUMMARY:
Approximately 10-27% of patients undergoing gynecologic surgeries develop a catheter associated urinary tract infection (CAUTI) in the post operatory period, as bladder catheterization is a common practice in gynecologic surgery. Cranberry products provide alternative means for preventing CAUTI and could result in decreased use of antimicrobials. In this pilot study we will enroll 200 women post gynecologic surgery and randomize them to take either cranberry powder capsules or placebo powder capsules. The low risk of harm associated with using cranberry to reduce UTI coupled with its potential benefit makes it a desirable intervention for the prevention of CAUTI. The conduct/ results of this pilot /feasibility study will prepare us for the conduct of a large scale clinical trial.

DETAILED DESCRIPTION:
Cranberry products prevent bacteria that cause UTI, especially Escherichia coli, from adhering to bladder cell wall thus preventing infection. Adherence of type 1 pili is inhibited by the fructose and of p pili by the proanthocyanidins present in cranberry.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting at the gynecology clinic for a pre-operatory visit
2. Ability to give informed consent
3. Willing to take cranberry capsules for up to 6 weeks
4. 18 of age or older

Exclusion Criteria:

1. Pregnancy
2. History of nephrolithiasis
3. History of allergy to cranberry
4. Patient on anticoagulant medicine to be re-started during the 4-6 weeks after surgery
5. Less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Foxman, PhD, Principal Investigator — University of Michigan
Locations (1):
- Urogynecology Clinic; University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Foxman B, Cronenwett AE, Spino C, Berger MB, Morgan DM. Cranberry juice capsules and urinary tract infection after surgery: results of a randomized trial. Am J Obstet Gynecol. 2015 Aug;213(2):194.e1-8. doi: 10.1016/j.ajog.2015.04.003. Epub 2015 Apr 13. PMID 25882919
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952
- [Derived] Manohar J, Hatt S, DeMarzo BB, Blostein F, Cronenwett AEW, Wu J, Lee KH, Foxman B. Profiles of the bacterial community in short-term indwelling urinary catheters by duration of catheterization and subsequent urinary tract infection. Am J Infect Control. 2020 Feb;48(2):178-183. doi: 10.1016/j.ajic.2019.08.005. Epub 2019 Sep 17. PMID 31540834

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at their preoperative appointment for gynecological surgery. At enrollment they completed a questionnaire about their history and signed an informed consent form. Participants were not assigned to a treatment arm until the day of their surgery.
Pre-assignment Details: If a participant's surgery was canceled or she failed to complete her enrollment questionnaire she was not assigned to a treatment arm.
  200 women were consented, 160 were randomly assigned to treatment (80 cranberry, 80 placebo).
Groups:
- Cranberry Capsules: Cranberry powder: 2 cranberry powder capsules twice a day
- Placebo: Placebo powder: 2 placebo powder capsules twice a day
Period: Overall Study
Arm/Group | Cranberry Capsules | Placebo
Started | 80 | 80
Completed | 67 | 63
Not Completed | 13 | 17
Not completed — Did not take a single dose | 6 | 4
Not completed — Lost to Follow-up | 3 | 4
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Protocol Violation | 2 | 3
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cranberry Capsules | Placebo | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Customized [Number; unit: participants]
  18 - 60 years | 47 | 48 | 95
  > 60 years | 33 | 32 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 80 | 160
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 75 | 77 | 152
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 69 | 72 | 141
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 80 | 80 | 160
Experienced a UTI in the past 12 mo [Number; unit: participants] — Participant has experienced UTI in the 12 months prior to her gynecologic surgery.
  participants | 18 | 19 | 37
Ever experienced UTI in life [Number; unit: participants] — Participant has experienced UTI at least once in her lifetime prior to her gynecologic surgery.
  participants | 49 | 50 | 99
Reasons for surgery [Number; unit: participants] — Categories are not mutually exclusive. Participants may have had more than one reason for surgery.
  participants
    Fibroids | 11 | 9 | 20
    Pelvic organ prolapse | 51 | 56 | 107
    Stress urinary incontinence | 21 | 23 | 44
    Chronic pelvic pain | 2 | 3 | 5
    Endometriosis | 0 | 2 | 2
    Abnormal uterine bleeding | 11 | 6 | 17
    Adnexal mass | 4 | 4 | 8
    Other | 9 | 18 | 27
Type of Surgery [Number; unit: participants] — Categories are not mutually exclusive; participants may have required more than one type of surgery.
  participants
    Urinary incontinence operation | 24 | 24 | 48
    Prolapse/reconstructive | 52 | 58 | 110
    Hysterectomy/other extirpative | 35 | 42 | 77
    Other | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Participants With Clinically-diagnosed and Treated UTI's.
Description: The primary endpoint was the number of participants who were clinically-diagnosed and treated for UTI whether or not results from a urine culture were available. All UTI's were confirmed via medical records.
Time Frame: From surgery to post-op visit, approximately 6 weeks post surgery
Population: Analysis was run on all 160 subjects that were ascribed to an arm of the study. Data were analyzed using an intent to treat protocol.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Cranberry Capsules | Placebo
Number analyzed (Participants) | 80 | 80
participants | 15 [11.71 to 28.66] | 30 [27.69 to 48.45]

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected beginning at time of randomization (admitted to surgery) and ended 30 days after their postoperative visit when study treatment ended (a total time period of 8-10 weeks).
Description: Adverse Events (AE) data were gathered via scheduled followup phone calls with participants and medical record review. UTI was an outcome and so was not reported as AE unless other pertinent symptoms occurred. Some severe AE's reported occurred before randomization but are reported here due to their severe nature.
Groups:
- Placebo Capsules: Placebo powder: 2 placebo powder capsules twice a day
Arm/Group | Cranberry Capsules | Placebo Capsules
Serious Adverse Events (participants affected / at risk) | 4/80 | 4/80
Other Adverse Events (participants affected / at risk) | 75/80 | 78/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cranberry Capsules (N=80) | Placebo Capsules (N=80)
Incarcerated hernia, small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolus in Right Lower Lobe (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Participant did not recover well from operation for incarcerated hernia so she has a CT scan that showed acute pulmonary embolus in the right lower lobe pulmonary artery branches.
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1) — hospital re-admission.
Chest pain secondary to reflux (GERD) (Gastrointestinal disorders) | 1 (1) | 0 (0) — The participant was admitted to the chest pain center in stable condition.
Right hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — hip repair previous to gynecological surgery and study drug.
Vertebral compression fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant said she had back pain and found out it was a fracture. She had a vertebroplasty compression. Participant said that the back pain went away 2 days after the procedure. She was given oxycontin and Flexeril
Altered mental status and progressive fatigue due to chronic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Participant told pups that she started feeling disoriented, tired and could not talk in the morning. She went to the hospital and was admitted for two days. She underwent a blood transfusion and received two pints of blood.
Transfusion related acute lung injury versus post operative pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — PARTICIPANT DID NOT TAKE STUDY DRUG. Participant was kept in the hospital after gynecologic because of transfusion related acute lung injury.
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Surgery was not performed and PARTICIPANT NEVER RECEIVED STUDY DRUG
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atypical migraine (Nervous system disorders) | 1 (1) | 0 (0) — While watching television she had a sudden headache 'all over' along with a sore feeling in both her eyes, as well as one bout of emesis. Headaches continued in the morning so she went to emergency dept. She does not have any other meningeal signs.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cranberry Capsules (N=80) | Placebo Capsules (N=80)
ABNORMAL LAB RESULTS (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
BLEEDING (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
BLOODY NOSE (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
BUMP-LEFT GROIN AREA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
EDEMA (ONE SPECIFIED AS BILATERAL) (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
ELEVATED CHOLESTEROL (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ELEVATED LABS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ELEVATED WHITE BLOOD CELL COUNT (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
LOW HEMATOCRIT LEVELS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SUBSTANCE EXPOSURE (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SUPERFICIAL PHLEBITIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
SWELLING (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
VAGINAL SPOTTING (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ABNORMAL ECG (Cardiac disorders) | 3 (3) | 7 (7)
ABNORMAL EKG (Cardiac disorders) | 1 (1) | 1 (1)
ANGINA (Cardiac disorders) | 1 (1) | 0 (0)
BLOOD PRESSURE PROBLEMS (Cardiac disorders) | 0 (0) | 1 (1)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC ABNORMALITIES (Cardiac disorders) | 0 (0) | 1 (1)
CHEST PAIN (Cardiac disorders) | 0 (0) | 1 (1)
HEART PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSION (Cardiac disorders) | 1 (1) | 2 (2)
T-WAVE ABNORMALITY, T WAVE INVERSIONS IN LEADS III AND AVF (Cardiac disorders) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1)
VESTIBULITIS (Ear and labyrinth disorders) | 1 (2) | 0 (0)
ELEVATED GLUCOSE (Endocrine disorders) | 1 (1) | 3 (3)
ELEVATED LABS (Endocrine disorders) | 1 (1) | 0 (0)
ELEVATED TSH LEVELS (Endocrine disorders) | 1 (1) | 0 (0)
PERIMENOPAUSAL SYNDROME (Endocrine disorders) | 0 (0) | 1 (1)
PRIMARY HYPERPARATHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
TENDERNESS IN AXILLA (Endocrine disorders) | 0 (0) | 1 (1)
TSH ELEVATED (Endocrine disorders) | 1 (1) | 0 (0)
VAGINAL ATROPHY (Endocrine disorders) | 1 (1) | 0 (0)
VASOMOTOR SYMPTOMS (Endocrine disorders) | 2 (2) | 8 (8)
VASOVAGAL EPISODE (Endocrine disorders) | 0 (0) | 1 (1)
BLURRED VISION (Eye disorders) | 1 (1) | 0 (0)
CATARACTS (Eye disorders) | 1 (1) | 0 (0)
CORNEAL ABRASION (Eye disorders) | 0 (0) | 2 (2)
DISLOCATED INTRAOCULAR LENS IN CAPSULAR BAG OS (Eye disorders) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 1 (1) | 0 (0)
EYE PAIN (Eye disorders) | 1 (1) | 0 (0)
POST PROCEDURE TENDERNESS (Eye disorders) | 0 (0) | 1 (1)
VISION CHANGES/PROBLEMS (Eye disorders) | 2 (2) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 2 (2)
ABDOMINAL SWELLING (Gastrointestinal disorders) | 1 (1) | 0 (0)
BLOATING (Gastrointestinal disorders) | 3 (3) | 2 (2)
BOWEL ISSUES (Gastrointestinal disorders) | 1 (1) | 11 (11)
C.DIFFICELE COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
CHANGE IN BOWEL MOVEMENTS (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 19 (19) | 13 (13)
CONSTIPATION AND OBSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
CRAMPING (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHEA AND CONSTIPATION (ALTERNATING) (Gastrointestinal disorders) | 0 (0) | 2 (2)
DIARRHEA/LOOSE STOOL (Gastrointestinal disorders) | 4 (5) | 1 (1)
DIARRHEA-C.DIFF (Gastrointestinal disorders) | 0 (0) | 1 (1)
DISCOLORED FECES (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
ELEVATED LIVER FUNCTION TESTS (Gastrointestinal disorders) | 2 (2) | 0 (0)
EMESIS AND/OR NAUSEA (Gastrointestinal disorders) | 17 (17) | 22 (22)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FECAL URGENCY (Gastrointestinal disorders) | 1 (1) | 0 (0)
GAS PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1)
GAS RETENTION (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTROENTERITIS (Gastrointestinal disorders) | 2 (2) | 7 (7)
GERD (Gastrointestinal disorders) | 0 (0) | 3 (3)
GI BACTERIAL OVERGROWTH (Gastrointestinal disorders) | 0 (0) | 1 (1)
GI ISSUES RELATED TO IBS (Gastrointestinal disorders) | 2 (2) | 0 (0)
HEARTBURN (Gastrointestinal disorders) | 1 (1) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (2) | 1 (1)
HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
LOOSE STOOLS AND LEAKAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
MEDICATION INTOLERANCE (Gastrointestinal disorders) | 1 (1) | 1 (1)
NAUSEA AND APPETITE CHANGES (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA AND DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
RBS (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL TENDERNESS (General disorders) | 0 (0) | 1 (1)
ABDOMINAL TINGLING (General disorders) | 0 (0) | 1 (1)
ALLERGY (General disorders) | 1 (1) | 0 (0)
APPETITE CHANGES (General disorders) | 0 (0) | 1 (1)
BLADDER PERFORATION INTRA-OPERATIVELY (General disorders) | 0 (0) | 1 (1)
BLEEDING (General disorders) | 1 (1) | 0 (0)
BOWEL DISCOMFORT (General disorders) | 0 (0) | 1 (1)
BUG BITE (General disorders) | 1 (1) | 0 (0)
BUTTOCKPAIN/LABIAL BURN (General disorders) | 1 (1) | 0 (0)
CHILLS (General disorders) | 0 (0) | 2 (2)
CHILLS, VASOMOTOR SYMPTOMS (General disorders) | 0 (0) | 1 (1)
CHRONIC ENDOMETRITIS (General disorders) | 1 (1) | 0 (0)
DIAGNOSIS OF METASTASIS OF COLON CANCER (General disorders) | 1 (1) | 0 (0)
DIFFICULT VOIDING DUE TO SWELLING (General disorders) | 1 (1) | 0 (0)
DIZZINESS (General disorders) | 0 (0) | 1 (1)
EXTENDED UVULAR/UVULAR IRRITATION (General disorders) | 0 (0) | 1 (1)
FATIGUE AND DISCOMFORT WITH MOVEMENT (General disorders) | 0 (0) | 1 (1)
FATIGUE OR DECREASED ENERGY LEVEL (General disorders) | 3 (3) | 3 (3)
FEVER (General disorders) | 0 (0) | 2 (2)
HEMATOMA (General disorders) | 0 (0) | 1 (1)
INCISION PAIN (General disorders) | 0 (0) | 1 (1)
INCISION SEEPAGE (General disorders) | 0 (0) | 1 (1)
LOW VITAMIN D LEVEL (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 0 (0) | 1 (1)
MIGRAINE (General disorders) | 1 (1) | 0 (0)
OSTEOPENIA (General disorders) | 0 (0) | 1 (1)
PAIN - POST OPERATIVE (General disorders) | 1 (1) | 2 (2)
PAIN - PUBIC (General disorders) | 0 (0) | 1 (1)
PAIN BY LEFT HIP (General disorders) | 1 (1) | 0 (0)
PAIN IN LOWER BACK (General disorders) | 1 (1) | 0 (0)
PAIN IN RIGHT LEG (General disorders) | 0 (0) | 1 (1)
PANCREATIC MASS (General disorders) | 0 (0) | 1 (1)
POST OP PAIN VERSUS NEUROLOGIC/ NEUROPATHIC PAIN (General disorders) | 1 (1) | 0 (0)
TEETH PAIN (General disorders) | 1 (1) | 0 (0)
URINARY RETENTION (General disorders) | 0 (0) | 1 (1)
VAGINAL BLEEDING (General disorders) | 3 (3) | 0 (0)
VAGINAL DISCHARGE (General disorders) | 0 (0) | 1 (1)
VAGINAL DISCOMFORT (General disorders) | 0 (0) | 1 (1)
VULVAR PRURITIS (General disorders) | 0 (0) | 1 (1)
WEIGHT GAIN (General disorders) | 1 (1) | 0 (0)
WEIGHT LOSS DUE TO LOSS OF APPETITE (General disorders) | 0 (0) | 1 (1)
COMMON COLD (Immune system disorders) | 0 (0) | 1 (1)
LOW GRADE FEVER (Immune system disorders) | 1 (1) | 0 (0)
SINUS ISSUES (Immune system disorders) | 0 (0) | 1 (1)
BODY SUBSTANCE EXPOSURE (Infections and infestations) | 0 (0) | 2 (2)
CHILLS (Infections and infestations) | 0 (0) | 1 (1)
COLD SYMPTOMS (Infections and infestations) | 1 (1) | 0 (0)
ELEVATED WBL (Infections and infestations) | 0 (0) | 1 (1)
INFECTION OF INCISION SITE (ONE SPECIFIED ERYTHEMA) (Infections and infestations) | 0 (0) | 1 (2)
ONCHOLISIS (Infections and infestations) | 1 (1) | 0 (0)
SINUS PROBLEMS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
VIRAL SYNDRONE (Infections and infestations) | 1 (1) | 0 (0)
YEAST VAGINITIS (Infections and infestations) | 5 (5) | 2 (2)
CYSTOTOMY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ABNORMAL LABS (Investigations) | 0 (0) | 1 (1)
DIFFICULTY EATING AND DRINKING/APPETITE CHANGES (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
ABDOMINAL PAIN/PRESSURE (Musculoskeletal and connective tissue disorders) | 4 (5) | 10 (10)
ACHY (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
BILATERAL KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BRUISING (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
BUTTOCK/HIP PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CRAMPING (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
HEADACHE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HIP FRACTURE (R GREATER TROCHOUTER AVULSION FRACTURE) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
INCISION PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
JAW NUMBNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
LOWER BACK PACK (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
LOWER QUADRANT DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LUMP IN LOWER ABDOMIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MILD CARPAL TUNNEL SYNDROME ON RIGHT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL PAIN DUE TO TRAUMA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN FORM DILATOR (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN ON RIGHT SIDE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN WITH ACTIVITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PAIN/PRESSURE/SORENESS (Musculoskeletal and connective tissue disorders) | 18 (19) | 16 (17)
PATELLOFEMORAL DEGENERATIVE JOINT DISEASE AND DEGENERATIVE TEAR POSTERIOR TORN LATERAL MENISCUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
POST OPERATIVE REPAIR (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PRESSURE ON LEFT SIDE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RECTAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
RECTAL INDURATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SUPRAPUBIC/PUBIC PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
UPPER BACK/NECK/SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)
VAGINAL AND URETHRAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
DIZZINESS AND RINGING IN EARS (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS/VERTIGO (Nervous system disorders) | 3 (3) | 2 (2)
FALL (Nervous system disorders) | 0 (0) | 1 (1)
FATIGUE (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 6 (6) | 5 (5)
LATERAL FEMORAL CUTANEOUS NERVE INJURY (Nervous system disorders) | 0 (0) | 1 (1)
LEFT NEUROPATHY DUE TO SURGICAL POSITIONING AND LENGTH OF CARE (Nervous system disorders) | 1 (1) | 0 (0)
LEG NUMBNESS (Nervous system disorders) | 1 (1) | 0 (0)
LIGHTHEADEDNESS (Nervous system disorders) | 3 (3) | 2 (2)
MEMORY ISSUES (Nervous system disorders) | 2 (2) | 0 (0)
MIGRAINES (Nervous system disorders) | 2 (2) | 0 (0)
NEUROLOGIC PARENTHESES (Nervous system disorders) | 1 (1) | 0 (0)
POST OPERATIVE PARESTHESIS (Nervous system disorders) | 0 (0) | 1 (1)
PUDENDAL NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
SLEEP APNEA-NEW DIAGNOSIS (Nervous system disorders) | 1 (1) | 0 (0)
SLEEP DIFFICULTIES (Nervous system disorders) | 0 (0) | 2 (3)
VAGAL REACTION (Nervous system disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0)
MOOD DISTURBANCE (Psychiatric disorders) | 1 (1) | 0 (0)
STRESS INDUCED FATIGUE (Psychiatric disorders) | 0 (0) | 1 (1)
ANION GAP METABOLIC ACIDOSIS WITH CONCOMITANT METABOLIC ALKALOSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
BLADDER ERYTHEMA (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER SPASMS (Renal and urinary disorders) | 3 (3) | 4 (4)
CATHETER DISCOMFORT (Renal and urinary disorders) | 1 (1) | 1 (1)
ELEVATED CREATININE LEVEL (Renal and urinary disorders) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 3 (3) | 1 (1)
PAIN (Renal and urinary disorders) | 0 (0) | 1 (1)
POST OPERATIVE HEALING (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 0 (0) | 1 (1)
URETHRAL PAIN (Renal and urinary disorders) | 0 (0) | 2 (2)
URINARY FREQUENCY (Renal and urinary disorders) | 3 (3) | 0 (0)
URINARY URGENCY AND FREQUENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 5 (5) | 6 (6)
URINARY ISSUES (Renal and urinary disorders) | 14 (14) | 22 (23)
URINARY RETENTION (Renal and urinary disorders) | 12 (12) | 14 (16)
UTI Symptoms (Renal and urinary disorders) | 0 (0) | 3 (4)
VAGINAL BLEEDING (Renal and urinary disorders) | 0 (0) | 1 (1)
ABNORMAL ULTRASOUND RESULTS -THICKENED ENDOMETRIAL STRIPE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
CRAMPING WITH MINSES (Reproductive system and breast disorders) | 1 (1) | 0 (0)
DYSPAREUNIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ENLARGED UTERUS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
FEELING OF FULLNESS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
INCREASED DISCOMFORT DURING MENSES (Reproductive system and breast disorders) | 0 (0) | 1 (1)
LABIAL EDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PAIN WITH INTERMITTENT SELF CATH (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PELVIC PAIN V. POST OP DISCONFORT (Reproductive system and breast disorders) | 1 (1) | 0 (0)
PERINAEAL PAIN IN THE INTROITAL REGION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PERINEAL DESCENT (Reproductive system and breast disorders) | 0 (0) | 1 (1)
SWELLING/IRRITION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
URINARY FREQUENCY (Reproductive system and breast disorders) | 0 (0) | 1 (1)
URINARY LEAKAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL BLEEDING (Reproductive system and breast disorders) | 13 (13) | 16 (16)
VAGINAL CHANGES (Reproductive system and breast disorders) | 3 (3) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 6 (6) | 6 (6)
VAGINAL INFECTION (Reproductive system and breast disorders) | 0 (0) | 4 (4)
VAGINAL IRRITATION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL PAN/PRESSURE (Reproductive system and breast disorders) | 2 (2) | 1 (1)
VULVAR PRURITUS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
ABNORMAL CHEST EXAM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
AIRWAY ISSUES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
COUGHING EPISODES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
DESATURATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
LUNG ISSUES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
MILD COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OBSTRUCTIVE SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PERSISTENT COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
POSTNASAL DRIP AND NASAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
SINUS SYMPTOMS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
UPPER RESPIRATORY INFECTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
ABDOMINAL SENSITIVITY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
AGGLUTINATION BETWEEN ANTERIOR AND POSTERIOR WALLS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
AIR POCKET UNDER SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
BENIGN LESION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
BRUISE (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
BRUISING (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HAIR LOSS (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
HERPES ZOSTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
INCISION ISSUES (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
KELOID (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
LICHENS SCLEROSIS FLARE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PRURITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SKIN NUMBNESS AND TINGLING (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SORE TEMPLE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
TISSUE BULGE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
WOUND INFECTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
YEAST INFECTIONS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
EMOTIONAL STRESS (Social circumstances) | 1 (1) | 0 (0)
ABDOMINAL PAIN POST OP (Surgical and medical procedures) | 1 (1) | 2 (2)
BOTHERSOME STITICHES (Surgical and medical procedures) | 0 (0) | 1 (1)
DENTAL EXTRACTION (Surgical and medical procedures) | 0 (0) | 1 (1)
EXTENSIVE ADHESIVE DISEASE (Surgical and medical procedures) | 1 (1) | 0 (0)
FATIGUE (Surgical and medical procedures) | 0 (0) | 1 (1)
GRANULATION (Surgical and medical procedures) | 0 (0) | 1 (1)
HEALING WOUND (Surgical and medical procedures) | 0 (0) | 1 (1)
HEMATOMA (Surgical and medical procedures) | 0 (0) | 1 (1)
INCISIONAL PAIN (Surgical and medical procedures) | 2 (2) | 0 (0)
PAIN/DISCOMFORT (Surgical and medical procedures) | 4 (6) | 6 (6)
POST OP SWELLING (Surgical and medical procedures) | 1 (1) | 0 (0)
POST SITE HERNIA (Surgical and medical procedures) | 1 (1) | 0 (0)
POSTOPERATIVE DIFFICULTIES (Surgical and medical procedures) | 0 (0) | 2 (2)
RIGHT BUTTOCK PAIN DUE TO SURGICAL PROCEDURE (Surgical and medical procedures) | 0 (0) | 1 (1)
SLING REVISION AND WOUND EXPLORATION SURGERY (Surgical and medical procedures) | 0 (0) | 1 (1)
SORE SPOT/SUTURE DISCOMFORT (Surgical and medical procedures) | 0 (0) | 1 (1)
SWELLING (Surgical and medical procedures) | 1 (1) | 0 (0)
VAGINAL BLEEDING POST OPERATIVELY (Surgical and medical procedures) | 1 (1) | 2 (2)
CHRONIC HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
DILATED TORTUOUS VESSELS IN THE RIGHT RETROPUBIC SPACE (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No